CLINICAL TRIAL: NCT04714502
Title: Verification of Biomarkers to Examine Neonatal Asphyxia-induced Hypoxic-ischemic Encephalopathy Study on Neuro-developmental Follow-up at 2 Years A Prospective Multicenter Observational Study for Development of a Diagnostic Test
Brief Title: Asphyxia Associated Metabolite Biomarker Investigation 2
Acronym: AAMBI2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: InfanDx AG (Industry)
Collaborators: Cukurova University (Other); University Children's Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: AAMBI2
Record Dates: First submitted 2021-01-13; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Birth Asphyxia
Keywords: biomarkers; asphyxia; Hypoxic ischemic encephalopathy
MeSH Terms: conditions — Asphyxia Neonatorum; Asphyxia; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants enrolled in AAMBI1

SUMMARY:
Follow-up of participants of AAMBI1 study at age of at least 2 years. AAMBI1(ClinicalTrials.gov ID: NCT03354208): Verification of biomarkers in a human population for their ability to diagnose the severity of neonatal asphyxia. These biomarkers linked to asphyxia have been identified in animal studies.

DETAILED DESCRIPTION:
Follow-Up on neuro-developmental status of Study participants of AAMBI1. AAMBI1(ClinicalTrials.gov ID: NCT03354208): The aim of the study is to verify the application of combinations of several laboratory parameters in early postnatal blood samples, for identification of infants, who will suffer from early abnormal neonatal neurological outcome, in a population at risk. The population at risk is defined as term and late preterm (>36 weeks of gestation) human infants following perinatal hypoxia-ischemia with or without postnatal resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Infants previously enrolled in the AAMBI1 study

Exclusion Criteria:

* Missing valid written informed parental consent

Ages: 22 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children, who had been enrolled in the AAMBI study immediately after birth because they had been suspected to be at risk for perinatal brain injury (hypoxic-ischemic encephalopathy, HIE) and/or evaluated for hypothermia therapy or because they had been enrolled in AAMBI as healthy controls (with adaptation disorder only).
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Participants with normal neuro-developmental status | up to 42 month age
  All infants with normal neuro-developmental status
Participants with potentially abnormal neuro-developmental status | up to 42 month age
  All infants who do not fulfill outcomes 1, 3 or 4
Participants with abnormal neuro-developmental status - HIE | up to 42 month age
  Presence of adverse 2 years neuro-developmental outcome likely attributable to perinatal hypoxic-ischemic brain injury
Participants with abnormal neuro-developmental status - non-HIE | up to 42 month age
  Presence of adverse 2 years neuro-developmental Outcome not attributable to perinatal hypoxic-ischemic brain injury

CONTACTS AND LOCATIONS:
Overall Officials: Ron Meyer, Study Director — InfanDx AG
Locations (4):
- Turkey (Türkiye) (4):
  - Turkey Cukurova University, Adana
  - University of Firat, Elâzığ
  - Özel Güngören Hastanesi, Istanbul
  - Mersin University School of Medicine, Mersin

IPD SHARING:
Plan to Share IPD: No